CLINICAL TRIAL: NCT04717778
Title: Comparison of Salivary pH After Consuming Milk of Origin Vegetable vs Cow's Milk in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Tecnologica de Mexico (Other)
Responsible Party: Principal Investigator, Annia Marisol Avalos Mejía, Principal Investigator, Universidad Tecnologica de Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-100
Record Dates: First submitted 2021-01-12; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: pH
MeSH Terms: interventions — Soy Milk

STUDY DESIGN:
Intervention Model Description: The study was carried out in 21 first grade primary school children, they were given 5 types of milk, each one was measured on different days (Monday cow's milk, Tuesday coconut milk, Wednesday almond milk, Thursday soy milk, Friday rice milk).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pH milk (Experimental): Group of children who were given the different types of milk and only the pH was measured
  Interventions: Dietary Supplement: Comparison of salivary pH after consuming milk of origin vegetable vs cow's milk

INTERVENTIONS:
Dietary Supplement: Comparison of salivary pH after consuming milk of origin vegetable vs cow's milk — They were given 5 types of milk, each one was measured on different days (Monday cow's milk, Tuesday coconut milk, Wednesday almond milk, Thursday soy milk, Friday rice milk).
  Other Names: cow´s milk, coconut milk, almond milk, soy milk and rice milk

SUMMARY:
The study was carried out in 21 first grade primary school children, 100% aged 6 years, 52.4% were female. They were given 5 types of milk, each one was measured on different days (Monday cow's milk, Tuesday coconut milk, Wednesday almond milk, Thursday soy milk, Friday rice milk)

DETAILED DESCRIPTION:
* The study was carried out in 21 first grade primary school children, 100% aged 6 years, 52.4% were female.
* The group was given a brushing technique using a model and 2 videos were shown to reinforce the brushing technique and explanation of what was going to be done in the study.
* Supervised tooth brushing was performed in a group of 5 people.
* They were given 5 types of milk, each one was measured on different days (Monday cow's milk, Tuesday coconut milk, Wednesday almond milk, Thursday soy milk, Friday rice milk).
* Each child was given 7 plastic cups each day and asked to pour their saliva into the cup when instructed.
* The samples were taken with pH indicator strips and the result was recorded in personalized tables.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls from 3 to 6 years

Exclusion Criteria

* Boys and girls with allergies
* Children with lactose intolerance

Elimination criteria:

- Boys and girls who do not want to participate at the time of the study

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Sociodemographic results | 1 hour the sociodemographic data of all the children were taken.
  The study was carried out in 21 first grade primary school children, 100% aged 6 years, 52.4% were female.
pH results | The average time of pH evaluation for each milk per child was an hour and a half.
  30 minutes after tooth brushing, each child was asked for the first saliva sample (basal pH measurement).
  After taking the basal pH, each child was given a glass with 50 ml of the milk to be measured.
  Saliva samples were measured with pH indicator strips and the result was recorded on custom charts.
  The pH was taken at 5, 10, 20, 30, 40 and 50 minutes.
  The normality distribution test (Shapiro-Wilk) was applied to the quantitative variables, with p = 0.0001, so that the data present a non-parametric or free distribution.
  To assess whether there were differences between the pH of the groups, the Kuskal-Wallis test was applied. For basal pH, p = 0.0001, therefore the null hypothesis is rejected and we conclude that the basal pH level is different in the five milks. Average basal pH:
  Rice milk 7 Cow milk 6.9 Almond milk 6.6 Soy milk 6.4 Coconut milk 6

CONTACTS AND LOCATIONS:
Overall Officials: Annia Avalos, Master, Principal Investigator — Universidad Tecnológica Centroamericana
Locations (1):
- UNITEC, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
We are working on the article to publish it and for the study to be available.

REFERENCES:
- [Background] Vanga SK, Raghavan V. How well do plant based alternatives fare nutritionally compared to cow's milk? J Food Sci Technol. 2018 Jan;55(1):10-20. doi: 10.1007/s13197-017-2915-y. Epub 2017 Nov 2. PMID 29358791
- [Background] Hettinga K, van Valenberg H, de Vries S, Boeren S, van Hooijdonk T, van Arendonk J, Vervoort J. The host defense proteome of human and bovine milk. PLoS One. 2011 Apr 27;6(4):e19433. doi: 10.1371/journal.pone.0019433. PMID 21556375
- [Background] Cuppari C, Manti S, Salpietro A, Dugo G, Gitto E, Arrigo T, Sturiale M, Salpietro C. ALMOND MILK: A POTENTIAL THERAPEUTIC WEAPON AGAINST COW'S MILK PROTEIN ALLERGY. J Biol Regul Homeost Agents. 2015 Apr-Jun;29(2 Suppl 1):8-12. PMID 26634581